CLINICAL TRIAL: NCT06585345
Title: Clinical Study on the Safety and Efficacy of CD7 CAR-T Cell in Patients With Relapsed/Refractory Acute Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The General Hospital of Western Theater Command (Other)
Collaborators: YakeBiotech Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHWesternTheaterCommand
Record Dates: First submitted 2024-07-07; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Acute-Leukemia
Keywords: Acute-Leukemia; Relapsed; Refractory
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): CD7 positive relapsed or refractory acute leukemia
  Interventions: Biological: CD7 CAR-T cell

INTERVENTIONS:
Biological: CD7 CAR-T cell — Split intravenous infusion of CD7 CAR-T cells [dose escalating infusion of (1-100)x10^6 CD7 CAR-T cells/kg]

SUMMARY:
Acute leukemia is a malignant clonal disease of hematopoietic stem cells. At present, the treatment for acute leukemia is relatively limited, and it is still based on high-intensity chemotherapy drug therapy and hematopoietic stem cell transplantation. The prognosis of recurrent and refractory acute leukemia is poor, and there is a lack of effective treatment plan. CD7 is a specific target on the surface of T cells, and CD7 CAR-T is expected to provide a new therapeutic path for patients with relapsed refractory acute leukemia.This is an open, single-arm, single-center, prospective clinical study. The main objective of the clinical study is to evaluate the clinical safety and tolerability of CD7 CAR-T in the treatment of acute leukemia.

DETAILED DESCRIPTION:
CD7 expression was determined by flow cytometry. After the target was determined, the subjects received the target dose of CD7 CAR-T from 1×105 to 1×108 /kg. Each subject will start with a low dose of 1×105/kg and if there are no significant side effects will be increased to the next dose until the maximum tolerated dose is reached. A variety of adverse events (including neurological events, hematological events, infections, and secondary tumors) will be collected from the time of infusion of CAR T cells to 24 months after infusion. To understand the complete response rate (CR) and partial response rate (PR) at 3 months; Recurrence rate, progression-free survival (PFS) and overall survival (OS) after 1 to 5 years of CD7 CAR-T reinfusion; The amount and duration of CD7 CAR-T in vivo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with acute leukemia.
2. Acute leukemia complex/refractory cases with poor response to conventional chemotherapy: 1) patients who did not achieve complete remission after 2 courses of treatment with standard induced remission regimen; 2) Recurrence within 6 months after the first remission; 3) Relapse 6 months after the first remission, but failure to be treated again with the original induced remission regimen; 4) Recurrent patients.
3. At least 2 weeks or 5 half-lives (whichever is shorter) from the start of preconditioning chemotherapy after prior systemic treatment, except for immune checkpoint inhibitors/agonists; Systemic immune checkpoint inhibitor/agonist treatment is at least 3 half-lives away from pre-treatment chemotherapy (e.g., ipilimumab, etc.).
4. Toxic reactions caused by previous antitumor therapy must be stabilized and returned to ≤ grade 1 (except for clinically insignificant toxicity, such as baldness).
5. Over 14 years old, under 65 years old.
6. Physical Strength score 0-3 (ECOG standard)
7. No obvious active infection or graft-versus-host disease
8. Expected survival ≥3 months
9. Adequate kidney, liver, lung and heart function, defined as:

   Creatinine clearance (estimated by Cockcroft Gault formula) > 60 mL/min; Serum ALT/AST ≤ 2.5 ULN; Total bilirubin ≤1.5 ULN, excluding subjects with Gilbert's syndrome; Cardiac ejection fraction ≥ 50%, echocardiography confirmed centropericardial effusion, and ECG showed no clinically significant abnormal findings.

   There was no clinically significant pleural effusion. Baseline blood oxygen saturation under indoor ventilation was > 92%.
10. The serum pregnancy test results of fertile women must be negative (women who have undergone surgical sterilization or at least 2 years after menopause are considered to be infertile).

Exclusion Criteria:

1. The subject has had other malignancies, non-melanoma skin tumors, carcinoma in situ (e.g. Cervix, bladder, breast), unless disease-free survival of at least 3 years
2. Presence or suspicion of uncontrollable fungal, bacterial, viral or other infections.
3. Known human immunodeficiency virus (HIV) infection
4. Known history of hepatitis B (HBsAg positive) or hepatitis C (HCV antibody positive). Subjects with latent or prehepatitis B infection (defined as HBcAb positive and HBsAg negative) can be enrolled only if PCR tests for HBV DNA are negative. In addition, these subjects were required to undergo a monthly PCR test for HBV DNA. Participants who are serologically positive for HCV antibodies can also be enrolled if their PCR test results for HCV RNA are negative.
5. Existing or past CNS disease, such as seizures, cerebrovascular ischemia/bleeding, dementia, cerebellar disease, or any CNS-related autoimmune disease
6. Subjects with severe heart disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months prior to screening, or any grade 3 (moderate) or 4 (severe) heart disease (according to the New York Heart Society Functional Grading Method NYHA) with lymphoma infiltrating the heart's atria or ventricles
7. A history of myocardial infarction, angioplasty or stent placement, unstable angina pectoris, or other clinically significant heart disease in the 12 months prior to enrollment
8. Emergency treatment is expected or likely to occur within 6 weeks due to rapid tumor progression (e.g. tumor mass compression)
9. Primary immune deficiency
10. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to enrollment
11. Any medical condition that may affect the evaluation of safety or efficacy
12. Have had severe rapid hypersensitivity reactions to any of the drugs to be used in this study
13. Administer live vaccine within ≤6 weeks prior to initiation of the pretreatment regimen
14. Pregnant or lactating female subjects
15. Male or female subjects who do not consent to effective contraception from the time they sign informed consent until 6 months after completing AT19 treatment
16. Subjects judged by the investigator had difficulty completing all visits or procedures required by the study protocol (including follow-up visits), or were not compliant enough to participate in the study
17. In the past 2 years, subjects have had other malignancies, non-melanoma skin tumors, carcinoma in situ (e.g. Cervix, bladder, breast), end-organ damage due to autoimmune diseases (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), or need to systematically administer immunosuppressive or other drugs for systemic disease control. Unless disease free survival of at least 3 years
18. Participate in other clinical experimenters during the same period

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 months
  Adverse events are evaluated with CTCAE V4.03
Overall response rate (ORR) | 24 months
  ORR includes CR, CRi, MLFS and PR. Complete remission (CR)#Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0x 10^9/L; platelet count >100x10^9/L. CR with incomplete hematologic recovery (CRi)#All CR criteria except for residual neutropenia (<1.0x10^9/L) or thrombocytopenia (<100x10^9/L). Morphologic leukemia-free state (MLFS): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required. Partial remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.

SECONDARY OUTCOMES:
Duration of overall response (DOR) | 24 months
  Duration of overall response will be assessed from the CAR-T cell infusion to progression, death or last follow-up
Progression-free survival(PFS) | 24 months
  PFS will be assessed from the CAR-T cell infusion to progression, death or last follow-up.
Overall survival(OS) | 24 months
  OS will be assessed from the CAR-T cell infusion to death or last follow-up

OTHER OUTCOMES:
the duration of CAR T-cells in vivo | 24 months
  the time of CAR-T cells' persistence in blood and the copies of CAR-T cells
CAR-T related cytokine expression | 24 months
  CAR-T related cytokine expression

CONTACTS AND LOCATIONS:
Overall Officials: Hai Yi, Ph.D, Principal Investigator — The General Hospital of Western Theater Command
Locations (1):
- The General Hospital of Western Theater Command, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT06585345/Prot_000.pdf